CLINICAL TRIAL: NCT01922479
Title: Pilot RAndomized Controlled Trial of FerrIC CarboxymaltosE in ASIAns With Heart Failure (the PRACTICE-ASIA-HF) Study
Brief Title: Pilot Study of Ferric Carboxymaltose to Treat Iron Deficiency in Asians With Heart Failure
Acronym: PRACTICEASIAHF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University Heart Centre, Singapore (Other); Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/00265; IMU/BFA/2012/12 (Other Grant/Funding Number: NUHS IMU Bridging Fund Award 2012)
Record Dates: First submitted 2013-08-11; First posted 2013-08-14 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Heart Failure; Anemia; Iron Deficiency
Keywords: Heart Failure; Anemia; Iron Deficiency; Ferric Carboxymaltose; Asian
MeSH Terms: conditions — Heart Failure; Anemia; Iron Deficiencies | interventions — ferric carboxymaltose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferric Carboxymaltose (Experimental): 1000mg intravenous Ferric Carboxymaltose, given as undiluted slow bolus injection over 15 minutes. Allowed to take concomitant oral iron supplements in usual clinical doses as prescribed clinically by attending physicians.
  Interventions: Drug: Ferric Carboxymaltose
- Placebo (Active Comparator): 20mls intravenous Normal Saline (0.9%), given as slow bolus injection over 15 minutes. Allowed to take oral iron supplements in usual clinical doses as prescribed clinically by attending physicians.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric Carboxymaltose — 1000mg intravenous Ferric Carboxymaltose, given as undiluted slow bolus injection over 15 minutes. Allowed to take concomitant oral iron supplements in usual clinical doses as prescribed clinically by attending physicians.
  Other Names: FerInject
  Arms: Ferric Carboxymaltose
Drug: Placebo — 20mls intravenous Normal Saline (0.9%), given as slow bolus injection over 15 minutes. Allowed to take concomitant oral iron supplements in usual clinical doses as prescribed clinically by attending physicians.
  Arms: Placebo

SUMMARY:
Heart failure (HF) is a major global public health issue which also affects Asia. Data from the National Registry of Disease in Singapore shows a 9.4% rise in HF admissions in public hospitals from 2008 to 2009 (4140 to 4530). Anaemia (low blood Haemoglobin level) is a common problem occurring in HF, ranging from 14% to 56% in outpatient registries and clinical trials. Anaemia exacerbates the basic symptoms of HF of dyspnea and exercise intolerance, thereby reducing quality of life (QoL). However, recent approaches aimed at improving and normalizing Haemoglobin have been unsuccessful.Novel approaches are required to address this problem. Iron deficiency (ID) is a well-understood cause of anaemia. ID without overt anaemia may be present in HF patients. A recent study by Jankowska et al published in 2010 of 546 HF patients showed a 37% prevalence of ID, regardless of Haemoglobin level. This was associated with worse outcomes including impaired exercise capacity. The presence of ID indicates a higher likelihood of deteriorating and dying early. A landmark study published in the New England Journal of Medicine (The Ferinject Assessment in Patients with Iron Deficiency and Chronic Heart Failure (FAIR-HF) study) showed that HF patients who were treated with IV iron in the form of Ferric Carboxymaltose (FCM) had better outcomes, including improved exercise capacity, overall function, and quality of life.

There is a lack of contemporary data on ID in HF patients in Asia, including data on treatment with this novel IV iron FCM.

Hypothesis We hypothesise that treating ID in HF patients in Asia using FCM will improve outcomes including exercise capacity, quality of life, overall functional status, and the need to be hospitalised for complications arising from HF.

DETAILED DESCRIPTION:
Heart failure (HF) is a major global public health issue which also affects Asia. Singapore National Registry of Disease data shows a 9.4% rise in public hospital HF admissions from 2008 to 2009 (4140 to 4530). Anaemia (low blood Haemoglobin level) is a common co-morbidity in HF, ranging from 14% to 56% in outpatient registries and clinical trials. Anaemia exacerbates the basic symptoms of HF of dyspnea and exercise intolerance, thereby reducing quality of life (QoL). However, recent approaches aimed at improving and normalizing Haemoglobin have been unsuccessful (STAMINA-HeFT, RED-HF).Novel approaches are required to address this problem. Iron deficiency (ID) is a well-understood cause of anaemia. ID without overt anaemia may be present in HF patients. The study by Jankowska (2010) of 546 systolic HF patients had a 37% prevalence of ID, regardless of Haemoglobin level. This was associated with reduced peak oxygen consumption, high ventilatory response, impaired exercise capacity, and depressive symptoms in HF patients. ID was a strong independent predictor of death, heart transplantation, and poor clinical outcome in chronic HF.The Ferinject Assessment in Patients with Iron Deficiency and Chronic Heart Failure (FAIR-HF) study showed significant improvement in 6MWT, NYHA class, and overall QoL score in HF patients treated with IV iron in the form of Ferric Carboxymaltose (FCM).Unpublished preliminary data from the ongoing Nation-wide Singapore study on Heart Failure (SHOP) indicates that the observed point prevalence of ID is approximately 60% with a significant and direct correlation with exercise performance.To date, no studies exist of FCM in an Asian HF population. We hypothesise that IV Iron repletion therapy using FCM in Asian patients with HF and ID will improve outcomes including exercise capacity (measured by 6MWT), quality of life (measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ amp; VAS), NYHA functional class, and rate of HF hospitalization.

Primary Aim To determine the effect of IV iron repletion therapy compared to placebo on exercise capacity change as assessed by the 6MWT at the 4th and 12th week after administration of IV FCM in subjects with recent acutely decompensated heart failure and iron deficiency.

Secondary Aims To assess the effect of IV FCM compared with placebo on change in QoL assessments (KCCQ amp; VAS).To assess the effect of IV FCM compared with placebo on change in NYHA Functional Class.To assess the effect of IV FCM compared with placebo on the rate of HF Hospitalization.To assess the safety and tolerability of IV FCM compared to placebo.

Hypothesis We hypothesise that IV Iron repletion therapy using FCM in patients with HF and ID will improve outcomes including exercise capacity (measured by 6MWT), quality of life (measured by KCCQ amp; VAS), NYHA functional class, and rate of HF hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for HF (regardless of LVEF)
* Capable of completing the 6MWT
* Screening TSAT <20%, Serum Ferritin <300 ng/mL and Hb≤14 g/dL
* At least 21 years of age
* Written informed consent.

Exclusion Criteria:

* Acute coronary syndrome
* Acute valvular heart dysfunction
* Known sensitivity to FCM
* IV iron therapy and/or blood transfusion in the 4 weeks prior to randomisation
* Body weight ≤35 kg
* Active bacterial infection
* Haemochromatosis or other iron storage disorder
* Serious medical condition, emergency condition, uncontrolled systemic disease or any other medical condition that, in the judgment of the Investigator, prohibits the patient from participating or potentially completing the study
* Planned participation in any other interventional study or having received trial medication in the context of a clinical trial within the last 4 weeks prior to participating in this trial.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in 6MWT distance over time | 12 weeks
  Assess the change in the patient's 6MWT distance over time, from baseline, at 4 weeks, and at 12 weeks.

SECONDARY OUTCOMES:
Change in QoL as assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ) and the Visual Analogue Scale (VAS). | 12 weeks
  Assess the change in the patient's QoL as assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ) and the Visual Analogue Scale (VAS) over time, from baseline, at 4 weeks, and at 12 weeks.
Change in NYHA Functional Class | 12 weeks
  Assess the change in the patient's NYHA Functional Class over time, from baseline, at 4 weeks, and at 12 weeks.
Rate of HF Hospitalisation | 12 weeks
  Assess the change in the patient's Rate of HF Hospitalisation over time, from baseline, at 4 weeks, and at 12 weeks.
Summary of any adverse events reported during the study | 12 weeks
  Assess any and all adverse events reported during the study, from baseline to 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn SP Lam, MBBS, MRCP (UK), Study Chair — National University Heart Centre, Singapore; Poh Shuan Daniel Yeo, MBBS, MRCP(UK), Principal Investigator — Tan Tock Seng Hospital; Tee Joo Yeo, MBBS, MRCP (UK), Principal Investigator — National University Heart Centre, Singapore
Locations (2):
- Singapore (2):
  - National University Heart Centre, Singapore, Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore, Singapore